CLINICAL TRIAL: NCT06547398
Title: Prostate Adaptive Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Collaborators: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prostate ART
Record Dates: First submitted 2024-07-25; First posted 2024-08-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to Adaptive radiotherapy or standard radiotherapy, 2:1 randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive radiotherapy +/- margin reduction (Active Comparator): Phase 1 and 2: Treating Radiation Therapists (RTs) on the treatment machine will review the treatment target and organs at risk contours that are automatically generated on the plan of the day. They will modify these safely, as required, and then also approve the computer generated re-plan of the day, within the bounds of departmental protocols and decision guides (RT led).
  Phase 2 only: Margin reduction facilitated by adaptive radiotherapy.
  Interventions: Radiation: Adaptive radiotherapy +/- Margin Reduction
- Standard radiotherapy (Active Comparator): Patients will receive standard image guided radiotherapy
  Interventions: Radiation: Image guided radiotherapy

INTERVENTIONS:
Radiation: Adaptive radiotherapy +/- Margin Reduction — Radiotherapy using adaptive technology to recontour and replan daily as required. Reductions in the PTV margin will also be introduced in the second phase of this study.
  Other Names: ART
  Arms: Adaptive radiotherapy +/- margin reduction
Radiation: Image guided radiotherapy — Standard radiation treatment used in the department of radiation oncology for prostate cancer
  Other Names: IGRT
  Arms: Standard radiotherapy

SUMMARY:
Prostate ART is a two phase study looking at using adaptive radiotherapy to help reduce toxicity for prostate cancer patients.

Adaptive radiotherapy is a new technology that provides the ability to account for daily changes in anatomy. Adaptive radiotherapy also provides a foundation for which radiotherapy margins might be safely reduced.

Phase 1 of this study is looking to see if a radiation therapist centred adaptive workflow can be implemented. If phase 1 of this study is safe and feasible, the study will proceed to phase 2.

Part 2 of the study looks at using adaptive technology to reduce radiation treatment margins. The primary aim of this study is to see whether margin reduced treatment using adaptive radiotherapy can reduce side effects for prostate cancer patients.

DETAILED DESCRIPTION:
Despite major technological advancements in the delivery of pelvic radiation therapy including the use of dynamic therapy, image guidance, integrated boosting and stereotactic techniques, toxicity from pelvic radiation remains a significant issue impacting on patient's quality of life and preventing the delivery of higher (and more curative) doses of radiation. Although evidence showed that adaptive radiotherapy demonstrating promising reduction of acute toxicity, the uptake of adaptive radiotherapy remains poor as adaptive radiation therapy is very labour intensive, time consuming and usually requires a radiation oncologist (RO) and Medical Physicist in attendance to review/modify target contours. These practices of daily multi-disciplinary team (MDT) in person attendance is not sustainable in the long term.

Since 2021, Royal North Shore Hospital has been treating patients with cancer in the pelvic with Adaptive Radiation Therapy (ART) and Radiation Therapists (RT) at the site have undergone a rigorous University based Advanced Practitioner training programme.

This study aims to evaluate RT-led ART in a randomised trial to assess the safety and feasibility of ART in a two stage phase 3 randomised controlled trial. If this study can prove safety and feasibility in the first phase, it will proceed to the second phase of the study which will look at using adaptive radiotherapy to safely reduce CTV and PTV margins.

The primary aim of the study will be to measure the difference in combined acute patient reported gastrointestinal (GI) and genitourinary (GU) toxicity between ART with margin reduction versus standard radiotherapy. Secondary aims will be to look at differences in biochemical failure, the time efficiency of ART, the radiation dosimetric differences between the treatment arms and patients' perception of ART.

ELIGIBILITY:
Inclusion Criteria:

1. - Age > 18
2. Biopsy proven prostate malignancy
3. Definitive treatment is radiotherapy to the prostate alone
4. ECOG performance status 0-2
5. Ability to understand and the willingness to sign an informed consent

Exclusion Criteria:

1. Hip prosthesis
2. Patient separation from prostate centre to skin edge > 24cm, measured on diagnostic scan-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male over 18 years old
Enrollment: 130 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety of Adaptive Radiation Therapy via Radiation Therapists-led* treatment delivery (CTV coverage) | 12 months
  A comparison of Clinical Target Volume (CTV) dose coverage will be performed.
  The CTV dose coverage must be equal or better in 90% of fractions for 90% of patients compared with the virtual image guided radiotherapy (IGRT) fraction. Dose coverage will be calculated as the percent of CTV receiving at least 95% of the prescribed dose (TD).
Safety of Adaptive Radiation Therapy via Radiation Therapists-led* treatment delivery (OAR DVH constraints) | 12 months
  A comparison of organ at risk (OAR) dose-volume histogram (DVH) constraints will be performed.
  The OAR DVH dose constraints must be equal or better in 90% of fractions for 90% of patients compared with the virtual image guided radiotherapy (IGRT) fraction.
Feasibility of ART via RT-led* treatment delivery | 12 months
  At least 90% of patients must have 90% of planned adaptive treatments successfully delivered in phase 1 of the study.
Acute patient reported toxicity | Within 90 days of patients completing treatment
  The study will measure the difference in patient reported combined maximum GU and GI toxicity (Grade 2 or higher) as per PRO-CTCAE between the two treatment arms.

SECONDARY OUTCOMES:
Acute clinician reported toxicity | Within 90 days of patients completing treatment
  The study will measure the difference in acute combined maximum GU and GI toxicity (Grade 2 or higher) grading between the two treatment arms as reported by clinicians using CTCAE v5.0
Late clinician reported toxicity | 5 years
  The study will measure the difference in late GU and GI toxicity (Grade 2 or higher) between the two treatment arms as reported by clinicians using CTCAE v5.0
Late patient reported toxicity | 5 years
  The study will measure the difference in patient reported late GU and GI toxicity (Grade 2 or higher) between the two treatment arms as per PRO-CTCAE.
Biochemical progression Free Survival | 3 and 5 years
  The rate of biochemical failure as defined as Nadir+2.0, commencement of ADT for relapse or evidence of disease recurrence on imaging
Time differences between treatment arms | 1 and 5 years
  The study will assess the average absolute treatment time difference per fraction for adaptive radiation therapy compared to prostate IGRT.
Radiation dosimetric differences between treatment arms | 1 and 5 years
  The study will evaluate the radiation dosimetric differences between treatment using ART and treatment using standard prostate IGRT
Patient reported attitudes and perceptions | 1 and 5 years
  The study will assess the patient experience with radiotherapy on a five item questionnaire that uses a five-point Likert-scale (ranging from strongly disagree to strongly agree). Differences in responses for each question between the arms will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Prof Kneebone, MBBS, Principal Investigator — Northern Sydney Local Health District
Locations (1):
- Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Only group data will be published.